CLINICAL TRIAL: NCT06375018
Title: Effect of the Diaphragm Stretching Technique on Symptomatology in Young Adults With Nonspecific Low Back Pain: Randomized Controlled Trial
Brief Title: Effect of the Diaphragm Stretching Technique on Nonspecific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Principal Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OST1_011
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Nonspecific Low Back Pain
Keywords: Diaphragm; Low Back Pain; Osteopathy; Osteopathic Medicine; Stretching Technique; Young Adults
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): After data collection, each volunteer will undergo a simulated technique within this group. The investigator will mimic the contacts of the phrenic nerve inhibition technique without applying traction or compression to the tissue, merely maintaining the contacts for the same duration as described in the technique performed in the experimental group, along with the same rest period afterward. Subsequently, new data will be collected following the simulated intervention.
  Interventions: Other: Placebo Technique
- Experimental group (Experimental): After collecting data from each volunteer, a Diaphragm Stretching technique will be administered to individuals in this group. The technique will be executed for a maximum duration of 4 minutes. Following the technique, volunteers will be required to rest for 5 minutes. Subsequently, another round of data collection will be conducted.
  Interventions: Other: Diaphragm Stretching

INTERVENTIONS:
Other: Placebo Technique — In the control group, manual contact will be carried out without any therapeutic intention. This contact will be maintained for the same period of time as the experimental group.
  Arms: Control group
Other: Diaphragm Stretching — The participant will be in supine position and the researcher will be at the headrest of the examination table, placing his hands on the lower costal margin. Superior direction traction is performed during inspiration, remaining during expiration. The procedure is repeated for a maximum period of 4 minutes.
  Arms: Experimental group

SUMMARY:
This study aims to analyze the efficacy of diaphragm stretching technique on symptomatology in young adults with nonspecific low back pain.

DETAILED DESCRIPTION:
Nonspecific low back pain occurs when there is an imbalance in the lower back between functional load and the ability to perform daily tasks. It is characterized as such when there is no specific and well-determined diagnosis and there are no structural changes.

The diaphragm and abdominal muscles together create a hydraulic effect in the abdominal cavity, which helps stabilize the spine, providing rigidity to the lumbar spine by increasing intra-abdominal pressure. Diaphragmatic changes in patients diagnosed with low back pain may contribute to the lack of spinal control activity through several mechanisms. Thus, it is concluded that the diaphragm is anatomically related to the lumbar spine, through its muscle fibers.

There are articles that relate the topic of low back pain with Osteopathic Manual Treatment, demonstrating that, despite this lack of scientific evidence, the results obtained at a clinical level are favorable.

This study aims to evaluate the effectiveness of diaphragm stretching techniques on symptoms experienced by young adults with non-specific low back pain.

In this study, the investigators will analyze the effects of the diaphragm stretching technique on the following variables: the sniff nasal inspiratory pressure test (SNIP test) , Visual Analogue Scale (VAS) score, the Schober test and measurement of the distance between the fingers and the ground during anterior flexion of the trunk, without flexion of the lower limbs (also known as the Finger Tip Test).

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific low back pain;
* Age between 18 and 30.

Exclusion Criteria:

* Serious cardiovascular and cardiorespiratory causes;
* Spinal pathologies and injuries to the lumbar spine;
* Cancer patients;
* Pacemaker or implant carriers;
* Pregnant women or volunteers suspected of being pregnant.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in level of inspiratory capacity immediately after intervention | Immediately after the intervention
  Assessment instruments to assess the degree of disability resulting from low back pain include the respiratory pressure meter.
Change in the level of disability derived from low back pain immediately after the intervention | Immediately after the intervention
  Assessment instruments to evaluate the degree of disability resulting from low back pain include the Visual Analogue Scale. In this scale, a higher score indicates a greater level of pain, correlating with a worse outcome. Conversely, a lower score indicates less pain, corresponding to a better outcome.
Change in the level of functionality of the lumbar spine immediately after the intervention | Immediately after the intervention
  Assessment instruments to assess the degree of disability resulting from low back pain include the Schober test.
Change in the level of functionality of the lumbar spine immediately after the intervention | Immediately after the intervention
  Assessment instruments to assess the degree of disability resulting from low back pain include the measurement of the distance from the hands to the floor after forward flexion of the trunk while standing with knee extension (also known as the Finger Tip Test).

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Porto
Locations (1):
- Escola Superior de Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Hodges PW, Eriksson AE, Shirley D, Gandevia SC. Intra-abdominal pressure increases stiffness of the lumbar spine. J Biomech. 2005 Sep;38(9):1873-80. doi: 10.1016/j.jbiomech.2004.08.016. PMID 16023475
- [Background] Hodges PW, Heijnen I, Gandevia SC. Postural activity of the diaphragm is reduced in humans when respiratory demand increases. J Physiol. 2001 Dec 15;537(Pt 3):999-1008. doi: 10.1111/j.1469-7793.2001.00999.x. PMID 11744772
- [Background] Bains KNS, Kashyap S, Lappin SL. Anatomy, Thorax: Diaphragm. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519558/ PMID 30137842
- [Background] Hodges PW, Cresswell AG, Daggfeldt K, Thorstensson A. In vivo measurement of the effect of intra-abdominal pressure on the human spine. J Biomech. 2001 Mar;34(3):347-53. doi: 10.1016/s0021-9290(00)00206-2. PMID 11182126
- [Background] Fernandez-Lopez I, Pena-Otero D, Atin-Arratibel MLA, Eguillor-Mutiloa M. Effects of Manual Therapy on the Diaphragm in the Musculoskeletal System: A Systematic Review. Arch Phys Med Rehabil. 2021 Dec;102(12):2402-2415. doi: 10.1016/j.apmr.2021.03.031. Epub 2021 Apr 29. PMID 33932362
- [Background] Finta R, Nagy E, Bender T. The effect of diaphragm training on lumbar stabilizer muscles: a new concept for improving segmental stability in the case of low back pain. J Pain Res. 2018 Nov 28;11:3031-3045. doi: 10.2147/JPR.S181610. eCollection 2018. PMID 30568484
- [Background] Fitting JW. Sniff nasal inspiratory pressure: simple or too simple? Eur Respir J. 2006 May;27(5):881-3. doi: 10.1183/09031936.06.00007906. No abstract available. PMID 16707389
- [Background] Grimstone SK, Hodges PW. Impaired postural compensation for respiration in people with recurrent low back pain. Exp Brain Res. 2003 Jul;151(2):218-24. doi: 10.1007/s00221-003-1433-5. Epub 2003 May 21. PMID 12759796
- [Background] Heritier F, Rahm F, Pasche P, Fitting JW. Sniff nasal inspiratory pressure. A noninvasive assessment of inspiratory muscle strength. Am J Respir Crit Care Med. 1994 Dec;150(6 Pt 1):1678-83. doi: 10.1164/ajrccm.150.6.7952632.
- [Background] Hershkovich O, Grevitt MP, Lotan R. Schober Test and Its Modifications Revisited-What Are We Actually Measuring? Computerized Tomography-Based Analysis. J Clin Med. 2022 Nov 22;11(23):6895. doi: 10.3390/jcm11236895. PMID 36498470
- [Background] Heuch I, Hagen K, Heuch I, Nygaard O, Zwart JA. The impact of body mass index on the prevalence of low back pain: the HUNT study. Spine (Phila Pa 1976). 2010 Apr 1;35(7):764-8. doi: 10.1097/BRS.0b013e3181ba1531. PMID 20228714
- [Background] Hides J, Gilmore C, Stanton W, Bohlscheid E. Multifidus size and symmetry among chronic LBP and healthy asymptomatic subjects. Man Ther. 2008 Feb;13(1):43-9. doi: 10.1016/j.math.2006.07.017. Epub 2006 Oct 27. PMID 17070721
- [Background] Hodges PW, Gandevia SC. Activation of the human diaphragm during a repetitive postural task. J Physiol. 2000 Jan 1;522 Pt 1(Pt 1):165-75. doi: 10.1111/j.1469-7793.2000.t01-1-00165.xm. PMID 10618161
- [Background] Hodges PW, Gandevia SC. Changes in intra-abdominal pressure during postural and respiratory activation of the human diaphragm. J Appl Physiol (1985). 2000 Sep;89(3):967-76. doi: 10.1152/jappl.2000.89.3.967. PMID 10956340
- [Background] Hodges PW, Cresswell AG, Daggfeldt K, Thorstensson A. Three dimensional preparatory trunk motion precedes asymmetrical upper limb movement. Gait Posture. 2000 Apr;11(2):92-101. doi: 10.1016/s0966-6362(99)00055-7. PMID 10899662
- [Background] Hodges PW, Gurfinkel VS, Brumagne S, Smith TC, Cordo PC. Coexistence of stability and mobility in postural control: evidence from postural compensation for respiration. Exp Brain Res. 2002 Jun;144(3):293-302. doi: 10.1007/s00221-002-1040-x. Epub 2002 Apr 13. PMID 12021811
- [Background] Hodges PW, van Dieen JH, Cholewicki J. Time to Reflect on the Role of Motor Control in Low Back Pain. J Orthop Sports Phys Ther. 2019 Jun;49(6):367-369. doi: 10.2519/jospt.2019.0104. PMID 31151378
- [Background] Iwai K, Nakazato K, Irie K, Fujimoto H, Nakajima H. Trunk muscle strength and disability level of low back pain in collegiate wrestlers. Med Sci Sports Exerc. 2004 Aug;36(8):1296-300. doi: 10.1249/01.mss.0000135791.27929.c1. PMID 15292735
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397
- [Background] Kocjan J, Adamek M, Gzik-Zroska B, Czyzewski D, Rydel M. Network of breathing. Multifunctional role of the diaphragm: a review. Adv Respir Med. 2017;85(4):224-232. doi: 10.5603/ARM.2017.0037. PMID 28871591
- [Background] Kolar P, Sulc J, Kyncl M, Sanda J, Neuwirth J, Bokarius AV, Kriz J, Kobesova A. Stabilizing function of the diaphragm: dynamic MRI and synchronized spirometric assessment. J Appl Physiol (1985). 2010 Oct;109(4):1064-71. doi: 10.1152/japplphysiol.01216.2009. Epub 2010 Aug 12. PMID 20705944
- [Background] Krismer M, van Tulder M; Low Back Pain Group of the Bone and Joint Health Strategies for Europe Project. Strategies for prevention and management of musculoskeletal conditions. Low back pain (non-specific). Best Pract Res Clin Rheumatol. 2007 Feb;21(1):77-91. doi: 10.1016/j.berh.2006.08.004. PMID 17350545
- [Background] Langevin HM, Stevens-Tuttle D, Fox JR, Badger GJ, Bouffard NA, Krag MH, Wu J, Henry SM. Ultrasound evidence of altered lumbar connective tissue structure in human subjects with chronic low back pain. BMC Musculoskelet Disord. 2009 Dec 3;10:151. doi: 10.1186/1471-2474-10-151. PMID 19958536
- [Background] Licciardone JC, Moore S, Fix K, Blair LG, Ta K. Osteopathic manipulative treatment of patients with chronic low back pain in the United States: a retrospective cohort study. J Osteopath Med. 2023 Feb 3;123(5):259-267. doi: 10.1515/jom-2022-0212. eCollection 2023 May 1. PMID 36732038
- [Background] Lizier DT, Perez MV, Sakata RK. Exercises for treatment of nonspecific low back pain. Rev Bras Anestesiol. 2012 Nov-Dec;62(6):838-46. doi: 10.1016/S0034-7094(12)70183-6. PMID 23176991
- [Background] Ludington E, Dexter F. Statistical analysis of total labor pain using the visual analog scale and application to studies of analgesic effectiveness during childbirth. Anesth Analg. 1998 Sep;87(3):723-7. doi: 10.1097/00000539-199809000-00045. No abstract available. PMID 9728862
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Marti-Salvador M, Hidalgo-Moreno L, Domenech-Fernandez J, Lison JF, Arguisuelas MD. Osteopathic Manipulative Treatment Including Specific Diaphragm Techniques Improves Pain and Disability in Chronic Nonspecific Low Back Pain: A Randomized Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1720-1729. doi: 10.1016/j.apmr.2018.04.022. Epub 2018 May 19. PMID 29787734
- [Background] Mrus JM, Yi MS, Freedberg KA, Wu AW, Zackin R, Gorski H, Tsevat J. Utilities derived from visual analog scale scores in patients with HIV/AIDS. Med Decis Making. 2003 Sep-Oct;23(5):414-21. doi: 10.1177/0272989X03256884. PMID 14570299
- [Background] Muehlbacher M, Nickel MK, Kettler C, Tritt K, Lahmann C, Leiberich PK, Nickel C, Krawczyk J, Mitterlehner FO, Rother WK, Loew TH, Kaplan P. Topiramate in treatment of patients with chronic low back pain: a randomized, double-blind, placebo-controlled study. Clin J Pain. 2006 Jul-Aug;22(6):526-31. doi: 10.1097/.ajp.0000192516.58578.a4. PMID 16788338
- [Background] Myles PS, Troedel S, Boquest M, Reeves M. The pain visual analog scale: is it linear or nonlinear? Anesth Analg. 1999 Dec;89(6):1517-20. doi: 10.1097/00000539-199912000-00038. PMID 10589640
- [Background] Nason LK, Walker CM, McNeeley MF, Burivong W, Fligner CL, Godwin JD. Imaging of the diaphragm: anatomy and function. Radiographics. 2012 Mar-Apr;32(2):E51-70. doi: 10.1148/rg.322115127. PMID 22411950
- [Background] Nava S, Ambrosino N, Crotti P, Fracchia C, Rampulla C. Recruitment of some respiratory muscles during three maximal inspiratory manoeuvres. Thorax. 1993 Jul;48(7):702-7. doi: 10.1136/thx.48.7.702. PMID 8153917
- [Background] Nguyen C, Boutron I, Zegarra-Parodi R, Baron G, Alami S, Sanchez K, Daste C, Boisson M, Fabre L, Krief P, Krief G, Lefevre-Colau MM, Rannou F. Effect of Osteopathic Manipulative Treatment vs Sham Treatment on Activity Limitations in Patients With Nonspecific Subacute and Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2021 May 1;181(5):620-630. doi: 10.1001/jamainternmed.2021.0005. PMID 33720272
- [Background] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Background] Perez AM, Fernandez-Carnero S, Sicilia-Gomez-de-Parada C, Cuenca-Zaldivar N, Naranjo-Cinto F, Pecos-Martin D, Gallego-Izquierdo T, Nunez-Nagy S. Diaphragmatic Activation Correlated with Lumbar Multifidus Muscles and Thoracolumbar Fascia by B-Mode and M-Mode Ultrasonography in Subjects with and without Non-Specific Low Back Pain: A Pilot Study. Medicina (Kaunas). 2023 Feb 8;59(2):315. doi: 10.3390/medicina59020315. PMID 36837516
- [Background] Romer LM, Polkey MI. Exercise-induced respiratory muscle fatigue: implications for performance. J Appl Physiol (1985). 2008 Mar;104(3):879-88. doi: 10.1152/japplphysiol.01157.2007. Epub 2007 Dec 20. PMID 18096752
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Stanton TR, Latimer J, Maher CG, Hancock MJ. How do we define the condition 'recurrent low back pain'? A systematic review. Eur Spine J. 2010 Apr;19(4):533-9. doi: 10.1007/s00586-009-1214-3. Epub 2009 Nov 18. PMID 19921522
- [Background] Stokes IA, Gardner-Morse MG, Henry SM. Intra-abdominal pressure and abdominal wall muscular function: Spinal unloading mechanism. Clin Biomech (Bristol). 2010 Nov;25(9):859-66. doi: 10.1016/j.clinbiomech.2010.06.018. Epub 2010 Jul 23. PMID 20655636
- [Background] Stokes M, Rankin G, Newham DJ. Ultrasound imaging of lumbar multifidus muscle: normal reference ranges for measurements and practical guidance on the technique. Man Ther. 2005 May;10(2):116-26. doi: 10.1016/j.math.2004.08.013. Epub 2004 Nov 18. PMID 15922232
- [Background] Uldry C, Fitting JW. Maximal values of sniff nasal inspiratory pressure in healthy subjects. Thorax. 1995 Apr;50(4):371-5. doi: 10.1136/thx.50.4.371. PMID 7785009
- [Background] van Middelkoop M, Rubinstein SM, Verhagen AP, Ostelo RW, Koes BW, van Tulder MW. Exercise therapy for chronic nonspecific low-back pain. Best Pract Res Clin Rheumatol. 2010 Apr;24(2):193-204. doi: 10.1016/j.berh.2010.01.002. PMID 20227641
- [Background] Verbeek JH, van der Weide WE, van Dijk FJ. Early occupational health management of patients with back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2002 Sep 1;27(17):1844-51; discussion 1851. doi: 10.1097/00007632-200209010-00006. PMID 12221346
- [Background] Vicente-Campos D, Sanchez-Jorge S, Terron-Manrique P, Guisard M, Collin M, Castano B, Rodriguez-Sanz D, Becerro-de-Bengoa-Vallejo R, Chicharro JL, Calvo-Lobo C. The Main Role of Diaphragm Muscle as a Mechanism of Hypopressive Abdominal Gymnastics to Improve Non-Specific Chronic Low Back Pain: A Randomized Controlled Trial. J Clin Med. 2021 Oct 27;10(21):4983. doi: 10.3390/jcm10214983. PMID 34768502
- [Background] Vleeming A, Schuenke MD, Danneels L, Willard FH. The functional coupling of the deep abdominal and paraspinal muscles: the effects of simulated paraspinal muscle contraction on force transfer to the middle and posterior layer of the thoracolumbar fascia. J Anat. 2014 Oct;225(4):447-62. doi: 10.1111/joa.12227. Epub 2014 Aug 20. PMID 25139243
- [Background] Vostatek P, Novak D, Rychnovsky T, Rychnovska S. Diaphragm postural function analysis using magnetic resonance imaging. PLoS One. 2013;8(3):e56724. doi: 10.1371/journal.pone.0056724. Epub 2013 Mar 14. PMID 23516397
- [Background] Wallden M. The diaphragm - More than an inspired design. J Bodyw Mov Ther. 2017 Apr;21(2):342-349. doi: 10.1016/j.jbmt.2017.03.013. Epub 2017 Apr 6. No abstract available. PMID 28532878
- [Background] Willard FH, Vleeming A, Schuenke MD, Danneels L, Schleip R. The thoracolumbar fascia: anatomy, function and clinical considerations. J Anat. 2012 Dec;221(6):507-36. doi: 10.1111/j.1469-7580.2012.01511.x. Epub 2012 May 27. PMID 22630613
- [Background] Winkelstein BA, Weinstein JN, DeLeo JA. The role of mechanical deformation in lumbar radiculopathy: an in vivo model. Spine (Phila Pa 1976). 2002 Jan 1;27(1):27-33. doi: 10.1097/00007632-200201010-00009. PMID 11805632